CLINICAL TRIAL: NCT02852317
Title: Urinary Markers of Detrusor Overactivity in Spina Bifida Patients
Acronym: BUHD-SPINA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC14_8805
Record Dates: First submitted 2016-07-19; First posted 2016-08-02 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2016-07

CONDITIONS: Spina Bifida; Multiple Sclerosis; Spinal Cord Injury; Overactive Bladder
MeSH Terms: conditions — Spinal Dysraphism; Multiple Sclerosis; Spinal Cord Injuries; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Spina bifida patient
- Patients with multiple sclerosis
- Patients with spinal cord injury
- Patients with overactive bladder

SUMMARY:
The purpose of this study is to assess diagnostic performance of urinary markers of detrusor overactivity (Nerve Growth Factor (NGF), Brain-Derived Neurotrophic Factor (BDNF), adenosine triphosphate (ATP), Prostaglandine E2) in detected high pressure bladder un spina bifida patients.

ELIGIBILITY:
Inclusion Criteria:

Study arm:

* Spina bifida patient
* Seen consecutively in outpatient clinics
* Age > 18 years-old

Control arm:

* Patients with multiple sclerosis or spinal cord injury or overactive bladder
* Seen consecutively in urodynamics
* with lower urinary tract symptoms
* Age > 18 years-old

Exclusion Criteria:

* Positive urine culture
* History of urologic neoplasms
* History of interstitial cystitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with an urodynamic examination scheduled
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Accuracy of urinary markers will be evaluated by area under the curve (AUC) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de Rennes, Rennes, France